CLINICAL TRIAL: NCT05631964
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics, and Initial Efficacy of BL-M07D1 for Injection in Patients With Locally Advanced or Metastatic Digestive Tract Tumors and Other Solid Tumors
Brief Title: Phase I Clinical Study of BL-M07D1 in Locally Advanced or Metastatic Digestive Tract Tumors and Other Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: SystImmune Inc. (Industry); Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-M07D1-102
Record Dates: First submitted 2022-11-13; First posted 2022-11-30 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced or Metastatic Digestive Tract Tumors; Other Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants receive BL-M07D1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-M07D1

INTERVENTIONS:
Drug: BL-M07D1 — Administration by intravenous infusion

SUMMARY:
Evaluation of BL-M07D1 for injection in Phase I clinical study of safety, tolerability, pharmacokinetic Characteristics, and initial efficacy in patients with locally advanced or metastatic digestive tract tumors and other solid tumors.

DETAILED DESCRIPTION:
Phase Ia: To observe the safety and tolerability of BL-M07D1 in patients with locally advanced or metastatic digestive tract tumors and other solid tumors, determine the MTD and DLT of BL-M07D1, and evaluate the pharmacokinetic characteristics and immunogenicity of BL-M07D1. Phase Ib: To further observe the safety and tolerability of BL-M07D1 at the Phase Ia recommended dose and determine RP2D. To evaluate the initial efficacy, pharmacokinetic characteristics and immunogenicity of BL-M07D1.

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent voluntarily and follow protocol requirements.
2. No gender limitation.
3. Age: ≥18 years and ≤75 years (phase Ia); ≥18 years old (phase Ib).
4. The expected survival time is ≥3 months.
5. Patients with locally advanced or metastatic HER2-positive/low-expression digestive tract tumors and other solid tumors that are not operable and have been confirmed by histopathology and/or cytology, have failed standard therapy, are not available for standard therapy, or are not currently applicable for standard therapy; HER2 positive: IHC 3+, or IHC 2+ and ISH positive; Low HER2 expression: IHC 2+ and ISH negative, or IHC 1+.
6. Agree to provide archived tumor tissue samples or fresh tissue samples from the primary or metastatic lesion within 2 years (to detect HER2 expression or amplification in tumor pathological tissue and explore its correlation with effectiveness indicators of BL-M07D1); If a subject is unable to provide a tumor tissue sample, he/she may be enrolled after an investigator's evaluation if other admission criteria are met.
7. There must be at least one measurable lesion that meets the RECIST v1.1 definition.
8. ECOG score 0 or 1.
9. The toxicity of previous antitumor therapy was restored to ≤1 as defined by NCI-CTCAE v5.0(except for asymptomatic laboratory abnormalities considered by the investigators, such as elevated ALP, hyperuricemia, and elevated blood glucose; Toxicities with no safety risk, such as hair loss, hyperpigmentation, grade 2 peripheral neurotoxicity, etc.).
10. No serious cardiac abnormality, left ventricular ejection fraction ≥50%.
11. The level of organ function must meet the following requirements and meet the following standards:

    1. Bone marrow function: absolute neutrophil count (ANC) ≥1.5×109/L, platelet count ≥100×109/L, hemoglobin ≥90 g/L;
    2. Liver function: total bilirubin (TBIL≤1.5 ULN), AST and ALT ≤2.5 ULN in patients without liver metastasis, AST and ALT ≤5.0 ULN in patients with liver metastasis;
    3. Kidney function: Creatinine (Cr) ≤1.5 ULN, or creatinine clearance (Ccr) ≥50 mL/min (based on Cockcroft and Gault formula).
12. Coagulation function: International Standardized ratio (INR) ≤1.5, and activated partial thrombin time (APTT) ≤1.5ULN.
13. Urine protein ≤2+ or ≤1000mg/24h.
14. Albumin ≥30 g/L.
15. A pregnancy test must be performed within 7 days of starting treatment for premenopausal women who are likely to have children, the serum/urine pregnancy must be negative, and the pregnancy must be non-lactation; All enrolled patients (male or female) should take adequate barrier contraception throughout the treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. Antitumor therapy such as chemotherapy, biotherapy, immunotherapy, radical radiotherapy, major surgery, targeted therapy (including small-molecule tyrosine kinase inhibitors) within 4 weeks prior to initial administration or within 5 half-lives, whichever is shorter; Mitomycin and nitrosourea were administered within 6 weeks before the first administration. Oral fluorouracil drugs such as Tizio, capecitabine, or palliative radiotherapy within 2 weeks prior to initial administration; Traditional Chinese medicines or proprietary Chinese medicines with anti-tumor indications should be administered within 2 weeks before the first administration.
2. Previously received ADC drug therapy with camptothecin derivatives (topoisomerase I inhibitors) as toxins (Phase Ib only).
3. History of severe heart disease, such as symptomatic congestive heart failure (CHF) ≥2 (CTCAE 5.0), New York Heart Society (NYHA) ≥2 heart failure, history of transmural myocardial infarction, unstable angina, etc.
4. Prolonged QT interval (QTcF > 450 msec in men or 470 msec in women), complete left bundle branch block, and degree III atrioventricular block.
5. Active autoimmune or inflammatory diseases, such as systemic lupus erythematosus, psoriasis requiring systemic treatment, rheumatoid arthritis, inflammatory bowel disease, and Hashimoto's thyroiditis, other than type I diabetes, hypothyroidism that can be controlled by alternative therapy alone, skin diseases that do not require systemic treatment (e.g., vitiligo, psoriasis).
6. Other malignancies developed within 3 years of enrollment, excluding:(1)radical cervical carcinoma in situ or non-melanoma skin cancer;(2)the second primary cancer that has been completely cured and no recurrence within 3 years;(3)The researchers believed that both primary cancers could benefit from this study;(4)The investigators have clearly ruled out which primary tumor source the metastases belong to.
7. Unstable thrombotic events such as deep vein thrombosis, arterial thrombosis, and pulmonary embolism requiring therapeutic intervention within 6 months prior to screening; Thrombus formation associated with infusion set is excluded.
8. The poorly controlled pericardial effusion, pleural effusion and abdominal effusion with clinical symptoms were not suitable for inclusion by the researchers.
9. Hypertension poorly controlled by antihypertensive medications (systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg).
10. According to CTCAE v5.0, patients were defined as ≥3 lung disease, ≥2 radiation lung disease, present or history of interstitial lung disease (ILD).
11. Patients who received lung radiation therapy within 6 months with total dose ≥30 Gy.
12. Patients with active central nervous system metastases. But the researchers believe that patients with stable brain parenchymal metastases can be included. The definition of stability should meet the following four requirements:

    1. Seizures-free status lasting > 12 weeks with or without antiepileptic medication;
    2. No need for glucocorticoids;
    3. Two consecutive MRI scans (scan interval at least 4 weeks) showed stable imaging status;
    4. Asymptomatic patients stable for more than 1 month after treatment.
13. Patients with a history of allergy to recombinant humanized antibodies or human and mouse chimeric antibodies or to any excipient component of BL-M07D1.
14. Previous recipients of organ transplantation or allogeneic hematopoietic stem cell transplantation (Allo-HSCT).
15. In previous treatment with anthracyclines, the equivalent cumulative dose of doxorubicin was greater than 360 mg/m2.
16. Human immunodeficiency virus antibody (HIVAb) positive, active tuberculosis, active hepatitis B virus infection (HBV-DNA copy number > lower limit of detection) or active hepatitis C virus infection (HCV antibody positive and HCV-RNA > lower limit of detection).
17. Active infections requiring systemic treatment, such as severe pneumonia, bacteremia, sepsis, etc.
18. Had participated in another clinical trial within 4 weeks prior to the first dose (counting from the time of the last dose).
19. A pregnant or nursing woman.
20. Other conditions included in this clinical trial were not considered appropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Dose Limited Toxicity (DLT) | Up to 21 days after the first dose
  The incidence and severity of adverse events (TEAE) during treatment were graded according to the National Cancer Institute Standard for Common Terminology for Adverse Events (NCI-CTCAE, v5.0).
Phase Ia: Maximum Tolerated Dose (MTD) | Up to 21 days after the first dose
  In the dose increment stage, the highest dose whose estimated DLT rate is closest to the target DLT rate but does not exceed the upper bound of the equivalent interval of DLT rate is selected as MTD.
Phase Ib: Recommended Dose for Phase II Clinical Studies (RP2D) | Up to 21 days after the first dose
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-M07D1.

SECONDARY OUTCOMES:
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B07D1 . The type, frequency and severity of TEAE will be evaluated during the treatment of BL-M07D1 .
Cmax | Up to 21 days after the first dose
  Maximum serum concentration (Cmax) of BL-M07D1 will be investigated.
Tmax | Up to 21 days after the first dose
  Time to maximum serum concentration (Tmax) of BL-M07D1 will be investigated.
T1/2 | Up to 21 days after the first dose
  Half-life (T1/2) of BL-M07D1 will be investigated.
AUC0-t | Up to 21 days after the first dose
  AUC0-t is defined as area under the serum concentration-time curve from time 0 to the time of the last measurable concentration.
CL(Clearance) | Up to 21 days after the first dose
  To study the serum clearance rate of BL-M07D1 per unit time.
Ctrough | Up to 21 days after the first dose
  Ctough is defined as the lowest serum concentration of BL-M07D1 prior to the next dose will be administered.
Anti-drug antibody (ADA) | Up to approximately 24 months
  Frequency and titer of anti-BL-M07D1 antibody (ADA) will be evaluated.
Phase Ib: Objective response rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Phase Ib: Disease control rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Phase Ib:Duration of response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Phase Ib: Progression-free survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of BL-B07D1 to the first date of either disease progression or death, whichever occurs first.
Phase Ib: Overall Survival(OS) | Up to approximately 24 months
  The time between the start of study medication and death.

CONTACTS AND LOCATIONS:
Overall Officials: Weijian Guo, PHD, Principal Investigator — Fudan University; Jian Zhang, PHD, Principal Investigator — Fudan University
Locations (1):
- Fudan University ShangHai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No